CLINICAL TRIAL: NCT03420456
Title: Transcranial Pulse Near-Infrared Light in Generalized Anxiety Disorder: a Placebo-Controlled Study (Lighten-GAD)
Brief Title: Transcranial Pulse Near-Infrared Light in Generalized Anxiety Disorder: a Placebo-Controlled Study
Acronym: Lighten-GAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funding for reasons unrelated to safety or efficacy
Sponsor: Massachusetts General Hospital (Other)
Collaborators: NYU Langone Health (Other); Cerebral Sciences LLC (Unknown)
Responsible Party: Principal Investigator, Paolo Cassano, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002231
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Pilot study
Masking Description: This is an open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Light Therapy (Experimental): Transcranial light therapy penetrates the skin and brain using light energy and the light energy may activate under-stimulated brain regions.
  Interventions: Device: Transcranial Light Therapy

INTERVENTIONS:
Device: Transcranial Light Therapy — Transcranial light therapy penetrates the skin and brain using light energy; this makes transcranial light therapy noninvasive. Transcranial light therapy may activate under-stimulated brain regions.
  Other Names: Low Level Laser-Light Therapy; Photobiomodulation

SUMMARY:
Transcranial Light Therapy involves non-invasive and invisible beams of light that increase energy metabolism in the brain. Transcranial light therapy has been found to promote brain metabolism which may help people with anxiety. The research team proposes a novel approach to treating anxiety by using transcranial light therapy.

DETAILED DESCRIPTION:
The purpose of this study is to see if using Transcranial Light Therapy (TLT), also called near- infrared light, helps improve symptoms of generalized anxiety disorder (GAD). Subjects will be randomized at a 1:2 ratio into 2 groups: pulse light (TLT) and sham. The sham group will be randomized after 8 weeks at a 1:1 ratio in to TLT and sham.

The study involves 1 screening visit which may last up to 3 hours, 16 weekly study visits, and one follow-up visit. There are 2 in-office treatment visits, during which a clinician applies transcranial light therapy to the participant's head for about 30 minutes. The other study visits involve assessments with a study clinician. The participants will administer the treatment once daily at home during the 16-week treatment period.

If a participant qualifies for the study, the study team assigns the participant by chance to receive either active transcranial light therapy or sham transcranial light therapy treatment. During sham transcranial light therapy visits, the transcranial light therapy device will not produce near infrared waves (e.g., light energy that cannot penetrate the skin and cranium). Participants have more than an equal chance of being assigned to the active transcranial light therapy or the sham transcranial light therapy over the course of the study. Neither the participant, nor the clinician, nor any research staff other than the study statistician will know which study group the participant belongs.

Participants are randomized a second time after 8-weeks in the study. If the participant were in the sham group the first 8-weeks, that participant may receive the active transcranial light therapy treatment after re-randomization. If the participant were already in the active transcranial light therapy group during the first 8-weeks the participant continues receiving the active treatment. All in all, participants have a 2 in 3 chance of receiving the active transcranial light therapy treatment at some point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age at screening will be between 18 and 70 years old (inclusive).
* Diagnosis of generalized anxiety disorder (MINI) - primary disorder
* CGI-S ≥4 or higher, i.e., "moderately anxious"
* Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms plus spermicide) if sexually active.
* Subject Informed Consent obtained in writing in compliance with local regulations prior to enrollment into this study.
* The subject is willing to participate in this study for at least 16 weeks.
* Subjects will need to be on stable dose(s) of anti-anxiety treatments (if taking any) for at least six weeks prior to enrollment.

Exclusion Criteria:

* The subject is pregnant or lactating.
* Structured psychotherapy focused on treating the subject's anxiety (i.e. CBT) and other alternative interventions for anxiety are permitted if started at least 8 weeks prior to the screening visit.
* Substance dependence or abuse in the past 3 months.
* History of a psychotic disorder or psychotic episode (current psychotic episode per MINI assessment).
* Bipolar affective disorder (per MINI assessment).
* Unstable medical illness, defined as any medical illness which is not well-controlled with standard-of-care medications (e.g., insulin for diabetes mellitus, HCTZ for hypertension).
* Active suicidal or homicidal ideation (both intention and plan are present), as determined by C-SSRS screening.
* Cognitive impairment (MOCA<21)
* The subject has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be in proximity to any of the procedure sites.
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)
* Recent history of stroke (90 days).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Structured Interview Guide for the Hamilton Anxiety Scale (SIGH-A) | 8 weeks - Sequential-parallel comparison design
  This instrument is completed by the clinician based on his/her assessment of the patient's anxiety symptoms, using a structured interview, specific instructions, and defined anchor points. Answers to the questions are rated on a scale of 0-4, with higher scores indicating more severe pathology. Scores range between 0 to 56; <17 indicates mild severity, 18-24 mild-to-moderate severity, and 25-30 moderate to severe.

SECONDARY OUTCOMES:
Clinical Global Impressions - Severity and Improvement (CGI-S, CGI-I) | 8 weeks - Sequential-parallel comparison design
  These two instruments are scored 1-7 by the clinician based on assessment of the subject's overall clinical status. They measure, based on history and scores on other instruments: (a) symptom severity (CGI-S) and (b) clinical improvement (CGI-I).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cassano, MD, Principal Investigator — Center for Anxiety and Traumatic Stress Disorders
Locations (1):
- Massachusetts General Hospital- Center for Anxiety and Traumatic Stress Disorders, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Personally unidentifiable information will be sent to Dr. Anastasia Ivanova, a privately contracted biostatistician form Chapel Hill North Carolina, for consultation on analyses. All information sent to Dr. Ivanova uses acrostics in place of personally identifiable information.